CLINICAL TRIAL: NCT04053465
Title: The Effect of Heat Acclimation on Repeated Bouts of Strenuous Heat Stress, Hand Cooling Efficacy, and the Maintenance Thereof.
Brief Title: Heat Acclimation, Hand Cooling Efficacy, and Adaptation Maintenance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Douglas J Casa, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H14-188
Record Dates: First submitted 2019-08-07; First posted 2019-08-12 (Actual); Results first posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Heat
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise in heat group (Experimental): Exercise in a hot environment
  Interventions: Other: Heat acclimation
- Exercise in cool group (Placebo Comparator): Exercise in a cool environment
  Interventions: Other: Exercise in a cool environment

INTERVENTIONS:
Other: Heat acclimation — 14 days of aerobic exercise in a hot environment
  Arms: Exercise in heat group
Other: Exercise in a cool environment — 14 days of aerobic exercise in a cool environment
  Arms: Exercise in cool group

SUMMARY:
This study had three aims:

1. To determine the impact of consecutive days of exercise on thermoregulation and cardiovascular strain.
2. To determine the efficacy of a hand cooling device to cool individuals throughout a heat acclimation period.
3. To assess the maintenance of thermoregulatory and cardiovascular adaptations derived from heat acclimation during a 25-day intermittent exercise-heat exposure protocol.

DETAILED DESCRIPTION:
Participants completed 14 days of exercise heat acclimation in either a hot or cool environment, followed by a heat or cool exercise exposure every 5th day for 25 days. Cardiovascular, thermoregulatory, and perceptual strain were measured throughout exercise each day. Hydration assessment and stress response via blood biomarkers were measured before and after exercise. Aerobic capacity was measured before and after heat acclimation as well as after the intermittent exercise-heat exposure. Hand cooling was implemented periodically during exercise-heat stress visits to determine cooling efficacy before and after heat acclimation.

ELIGIBILITY:
Inclusion Criteria:

* no chronic health problems
* no previous history of exertional heat stroke within the past 3 years
* no history of cardiovascular, metabolic or respiratory disease
* no current musculoskeletal injury that limits physical activity

Exclusion Criteria:

* women
* exercise less than once per week
* VO2max < 45 ml/kg/min

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2015-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas J Casa, PhD, Principal Investigator — University of Connecticut

IPD SHARING:
Plan to Share IPD: No
Aggregate data can be shared upon request.

REFERENCES:
- [Derived] Pryor RR, Pryor JL, Vandermark LW, Adams EL, Brodeur RM, Armstrong LE, Lee EC, Maresh CM, Casa DJ. Short term heat acclimation reduces heat strain during a first, but not second, consecutive exercise-heat exposure. J Sci Med Sport. 2021 Aug;24(8):768-773. doi: 10.1016/j.jsams.2021.03.020. Epub 2021 Apr 6. PMID 33846088

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were excluded if they did not reach the aerobic fitness criteria or if there were foreseen scheduling conflicts.
Period: Overall Study
Arm/Group | Exercise in Heat Group | Exercise in Cool Group
Started | 22 | 12
Completed | 18 | 8
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise in Heat Group | Exercise in Cool Group | Total
Number analyzed (Participants) | 22 | 12 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 12 | 34
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 22 | 12 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 12 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 12 | 34
VO2max [Mean (Standard Deviation); unit: mL/kg/min] | 53.5 (1.7) | 56.9 (2.2) | 54.6 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Internal Body Temperature
Description: Rectal temperature was assessed five days following measurement at baseline.
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: degrees Celcius
Arm/Group | Exercise in Heat Group | Exercise in Cool Group
Number analyzed (Participants) | 22 | 12
degrees Celcius | 39.6 (0.47) | 38.2 (0.30)

2. Secondary Outcome: Heart Rate
Description: Heart rate was assessed five days following baseline.
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Exercise in Heat Group | Exercise in Cool Group
Number analyzed (Participants) | 22 | 12
beats per minute | 178 (17) | 173 (4)

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Exercise in Heat Group | Exercise in Cool Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/12
Other Adverse Events (participants affected / at risk) | 0/22 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes